CLINICAL TRIAL: NCT07227948
Title: Repurposing Semaglutide for the Treatment of Cocaine Use Disorder: a Pilot Mechanistic Study
Brief Title: Repurposing Semaglutide for the Treatment of Cocaine Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Luba Yammine, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-25-0412; R01DA062720-01 (NIH)
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cocaine Use Disorder
Keywords: semaglutide; GLP-1 agonist; cocaine addiction
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — semaglutide; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental)
  Interventions: Drug: Semaglutide; Behavioral: cognitive behavioral therapy (CBT).
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Behavioral: cognitive behavioral therapy (CBT).

INTERVENTIONS:
Drug: Semaglutide — Participants will receive 14 weekly injections administered subcutaneously. Semaglutide will be initiated at a dose of 0.25 mg once weekly. After 4 weeks, the dose will be increased to 0.5 mg once weekly for an additional 4 weeks. Thereafter, the dose will be increased to 1 mg once weekly for 6 weeks
  Arms: Semaglutide
Drug: Placebo — Sterile saline (0.9%) will serve as the placebo for semaglutide and will be administered subcutaneously once-weekly for 14 weeks. The placebo will be administered in the same blinded manner as semaglutide and will be volume-matched.
  Arms: Placebo
Behavioral: cognitive behavioral therapy (CBT). — Participants will receive fourteen weekly 1-hour sessions of individual cognitive behavioral therapy (CBT), an evidence-based behavioral therapy platform for evaluating pharmacotherapy for CUD. CBT focuses on (1) identifying situations that precipitate drug use and (2) preventing relapse by teaching cognitive and behavioral skills to reduce risk.

SUMMARY:
The purpose of this study is to evaluate semaglutide, a glucagon-like peptide-1 receptor agonist (GLP-1RA), in combination with cognitive behavioral therapy (CBT) for the treatment of cocaine use disorder (CUD).

DETAILED DESCRIPTION:
The United States is facing a resurgence in cocaine use and cocaine-related mortality. Despite the significant public health burden, there are no FDA-approved pharmacotherapies for CUD, and existing behavioral interventions, such as cognitive behavioral therapy (CBT), demonstrate only modest efficacy when used alone. Identifying pharmacological agents that can enhance the effectiveness of behavioral treatments remains a critical public health priority.

One particularly promising class of medications for CUD is glucagon-like peptide-1 receptor agonists (GLP-1RA). These agents are widely used to treat type 2 diabetes and obesity due to their ability to regulate blood glucose and support metabolic health. Importantly, GLP-1 receptors are expressed in brain regions involved in reward processing and hedonic behavior. Consistent with this, animal studies have shown that GLP-1RAs reduce the rewarding and reinforcing effects of various addictive substances, including cocaine. If similar effects are observed in humans, GLP-1RAs may improve treatment outcomes by directly reducing the motivational salience of cocaine and its cues, and/or by enhancing responsiveness to behavioral therapies such as CBT.

The primary objective of this trial is to provide proof-of-concept evidence for the use of a GLP-1RA semaglutide as a treatment for CUD. The study hypothesizes that semaglutide will modulate three key reward-related target mechanisms underlying cocaine use: (1) motivational relevance of cocaine cues, assessed via event-related potentials (ERPs); (2) cocaine valuation, measured by behavioral economic demand for cocaine; and (3) subjective experience of craving. These mechanisms will be evaluated using a multimodal approach - neurophysiological, behavioral, and self-report - within a framework of a randomized clinical trial. In addition to assessing changes in the proposed target mechanisms, the study will evaluate the impact of semaglutide on cocaine use.

This project addresses the urgent need to explore novel pharmacological targets using an experimental therapeutics framework and has the potential to accelerate the development of effective treatments for CUD. If successful, the findings will support a fully powered efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent before any study-related activity, willing to comply with all study procedures, and be available for the duration of the study.
* Meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM 5) diagnostic criteria for CUD and report recent cocaine use (verified by at least one positive urine drug screen (UDS) for the cocaine metabolite benzoylecgonine (BE), during intake).
* Have body mass index (BMI) of ≥25 kg/m2
* Agree (if the participant is female and of child-bearing potential) to use effective contraceptive methods, unless the participant's male partner(s) is surgically sterile (underwent vasectomy). Acceptable contraceptives include oral contraceptives, contraceptive sponge, patch, double barrier (diaphragm/spermicidal or condom/spermicidal), intrauterine contraceptive system, etonogestrel implant, medroxyprogesterone acetate contraceptive injection, complete abstinence from sexual intercourse, and/or hormonal vaginal ring. Contraceptive measures sold for emergency use after unprotected sex are not acceptable methods for routine use. Women of child-bearing potential must provide negative urine pregnancy test prior to randomization. Note: A woman is considered fertile (of childbearing potential) following menarche and until becoming postmenopausal unless permanently sterile. Women in the following categories are not considered a woman of childbearing potential: premenarcheal, premenopausal female with one of the following: documented hysterectomy, documented bilateral salpingectomy, documented bilateral oophorectomy. Postmenopausal female is defined as no menses for 12 months without an alternative medical cause. Females on HRT and whose menopausal status is in doubt will be required to use one of the nonhormonal highly effective contraception methods if they wish to continue their hormone replacement therapy (HRT) during the trial.
* Have a medical and psychiatric history and a brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the Study Physician and the Principal Investigator.
* Be able to provide the names of at least 2 persons who can consistently locate their whereabouts.

Exclusion Criteria:

Medical Exclusions

* Personal or first-degree relative(s) history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2).
* History or presence of chronic pancreatitis or recent acute pancreatitis.
* Type 1 or type 2 diabetes mellitus (previously diagnosed or indicated by HbA1C ≥48 mol/mol (6.5%) as measured at screening).
* Severe gastrointestinal disease (i.e., severe gastroparesis).
* History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed.
* History of severe cardiovascular disease.
* History of retinopathy.
* Systolic blood pressure (SBP) >180 mmHg and/or diastolic blood pressure (DBP) >105 mmHg)
* End stage renal disease (ESRD, previously diagnosed or indicated by estimated glomerular filtration rate (eGFR) value of eGFR < 15 ml/min/1.73 m2 at screening).
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥3 times the upper limit of normal range at screening.
* Known or suspected hypersensitivity to semaglutide, excipients, or related products.
* History of seizure or elevated risk of seizure.
* Women who are currently pregnant, or plan to become pregnant, or lactating, or of childbearing potential and are not using medically accepted forms of contraception
* Have any medical illness or condition which in the opinion of the PI and/or the Study Physician would preclude safe and/or successful completion of the study.
* Any foreseeable procedure requiring general anesthesia or deep sedation.

Psychiatric/Substance Use Exclusions

* Current ≥ moderate substance use disorder aside from alcohol, nicotine, or marijuana, or a Substance Use Disorder (SUD) requiring medical detoxification (e.g., alcohol, opioid, benzodiazepine)
* Current or recent suicidal ideation.
* Homicidal ideation that requires immediate attention.
* Have any psychiatric illness or condition which in the opinion of the PI and/or the Study Physician would preclude safe and/or successful completion of the study.

Weight-Related Exclusions

* Gained/lost ≥4.5 kg (10 lb.) over the past 6 months (prior to screening).
* Uncontrolled thyroid disease at screening

Medication-Related Exclusions

* Currently using sincalide, sulfonylureas, insulin and insulin products, or medication used for weight management (i.e., orlistat, naltrexone-bupropion, liraglutide, semaglutide, tirzepatide, phentermine, topiramate, benzphetamine, diethylpropion, phendimetrazine).
* Any otherwise not specified concomitant medication that could compromise participant safety or treatment in the opinion of the Study Physician and/or the PIs.

General Exclusions

* Current, anticipated, or pending enrollment in another addiction treatment program and/or research study that could potentially affect participant safety and/or the study data/design as determined by the Principal Investigator and/or Study Physician.
* Not planning to live in the area for the duration of the trial.
* Surgery scheduled for the duration of the trial, except for minor surgical procedures, in the opinion of the PI and/or the Study Physician.
* Unable to communicate (read, write, and speak) fluently in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2029-01-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Amplitude of the Late Positive Potential (LPP) in microvolts in response to visual stimuli on the Picture Viewing Task. | End of Treatment (Week 15)
  EEG will be recorded during a passive picture viewing presentation that will include cocaine-related, neutral, and nondrug-related pleasant and unpleasant images. For each participant, the amplitude of the LPP component will be calculated separately for each picture category and used to evaluate the motivational relevance of the images.LPP amplitude reflects the motivational relevance of visual stimuli, with larger amplitudes indicating greater motivational salience.
Intensity of demand as assessed by the amount of cocaine purchased and consumed as assessed by cocaine purchasing task | End of Treatment (Week 15)
  Participants will complete the hypothetical Cocaine Purchasing Task, in which they report the amount of cocaine they would purchase and use at escalating price levels. Demand curve metrics (Intensity, Omax, Pmax, and Elasticity) will be calculated to quantify the relative reinforcing value and motivation to obtain cocaine. Lower demand values indicate reduced motivation for cocaine.
Cocaine craving as assessed by the score on the Cocaine Cravings Questionnaire | End of Treatment (Week 15)
  Cocaine craving will be assessed using a 10-item self-report questionnaire. Each item is rated on a 5-point Likert scale from 1 = Strongly Disagree to 5 = Strongly Agree. The total craving score is calculated as the mean of all item responses, with higher scores indicating greater craving intensity.
Proportion of cocaine negative urine drug screens (UDS) during the final two weeks of treatment | From Week 13 to Week 14
  Use of cocaine at the end of treatment

SECONDARY OUTCOMES:
Treatment response as a dichotomous outcome during the last two weeks of treatment | From Week 13 to Week 14
  Defined as at least three cocaine-negative urine drug screens (UDS) during the last two weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Luba Yammine, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No